CLINICAL TRIAL: NCT04489264
Title: A Prospective Study of Consolidative Autologous Stem Cell Transplantation After First-line Therapy in Peripheral T Cell Lymphoma
Brief Title: The Role of Consolidative Autologous Stem Cell Transplantation After First-line Therapy in Peripheral T Cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Party secretary of Cancer Hospital of Peking University, Director of Internal Medicine, Peking University
Other Study IDs: ASCT for PTCL
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Autologous Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Transplantation, Autologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASCT group: patients who achieved CR or PR after 6-8 cycles first-line therapy receive ASCT as consolidation therapy
  Interventions: Drug: Transplant, Autologous
- Observation group: patients who achieved CR or PR after 6-8 cycles first-line therapy finish their therapy and go into follow-up

INTERVENTIONS:
Drug: Transplant, Autologous — high dose chemotherapy followed by autologous stem cell transplantation
  Groups: ASCT group

SUMMARY:
The role of autologous stem cell transplantation (ASCT) in the first remission (CR1 & PR1) of peripheral T-cell lymphomas (PTCLs) is not well defined. This study analyzed the impact of ASCT on the clinical outcomes of patients with newly diagnosed PTCL in CR1 and PR1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed pathological diagnosis of aggressive PTCL
* Age 18-65 years old
* Achieving CR or PR after first-line therapy

Exclusion Criteria:

* Subtypes with a more indolent course, including precursor T/natural killer neoplasms, T-cell large granular lymphocytic leukemia, mycosis fungoides other than transformed mycosis fungoides, Sézary syndrome, and primary cutaneous CD30-positive disorders.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: lymphoma patients in several hospitals in China
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2-year PFS

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, Dr., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No